CLINICAL TRIAL: NCT04644640
Title: Telerehabilitation Following Meniscectomy: A Randomized Clinical Trial
Brief Title: Telerehabilitation Following Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-01584
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Meniscectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Active Comparator)
  Interventions: Other: Telerehabilitation Therapy
- In-Person Rehabilitation (Active Comparator)
  Interventions: Other: In-person Rehabilitation Therapy

INTERVENTIONS:
Other: Telerehabilitation Therapy — Rehabilitation services will be dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information - range of motion exercises for the knee, proprioception and balance training
  Arms: Telerehabilitation
Other: In-person Rehabilitation Therapy — Range of motion exercises for the knee, proprioception and balance training
  Arms: In-Person Rehabilitation

SUMMARY:
Telerehabilitation is a form of tele-treatment in which rehabilitation services are dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information. Since telerehabilitation was found to be equally effective as conventional therapy, it was being practiced even before the COVID times, however it was truly valuable during the lockdown. The advantages of telerehabilitation include reducing unnecessary travel to the hospital and person to person contact while maintaining social distancing. While some of the patients are truly staying at remote areas, others are unable to manage travel in the lockdown period. Telemedicine offers the opportunity to deliver rehabilitative services in the patients' home, closing geographic, physical, and motivational gaps. Punctuality on either side is also assured since the travel times are saved on both the ends.

The purpose of the proposed study is to evaluate telerehabilitation vs in-person rehabilitation following Meniscectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for meniscectomy
* Age 18-75
* Ability to comply with a standardized postoperative protocol
* Willing and able to provide consent

Exclusion Criteria:

* Pregnant patient
* Age >75 years, or < 18
* Previous knee surgery
* Unable to speak English or perform informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Score | up to 1 year post-op
  VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The total score ranges from 0-10. The higher the score, the worse the pain.
International Knee Documentation Committee (IKDC) Score | up to 1 year post-op
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to kirk.campbell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.